CLINICAL TRIAL: NCT06439524
Title: The Effect of Medical Management Following Excisional Surgery for Endometriosis: A Randomized Controlled Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Main Line Health (Other)
Collaborators: Pfizer (Industry); Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2024-02-29; First posted 2024-06-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — relugolix; Estradiol; Norethindrone Acetate

STUDY DESIGN:
Intervention Model Description: The design of this study will be an unblinded randomized controlled trial of medical suppression with once daily Relugolix combination therapy (Rel-CT) following excisional surgery for endometriosis performed by high volume minimally invasive gynecologic surgeons. Researchers will use descriptive statistics to compare the demographics and clinical characteristics of the groups with chi-square and two-sample t-tests. The median differences in EHP-30 from baseline to 6 months will be compared between groups with Mann Whitney U test. The 95% confidence interval of the difference between group medians will be used to measure superiority.
Masking Description: Participants and providers will know if participants are assigned to the treatment arm to take Rel-CT or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rel-CT (Active Comparator): 40 mg relugolix, 1 mg estradiol, 0.5 mg norethindrone acetate, one tablet daily for 6 months
  Interventions: Drug: 40 mg relugolix, 1 mg estradiol, 0.5 mg norethindrone acetate
- no study drug (No Intervention): no study drug

INTERVENTIONS:
Drug: 40 mg relugolix, 1 mg estradiol, 0.5 mg norethindrone acetate — if randomized to study drug, participants will take one tablet Rel-CT daily following excisional surgery for endometriosis
  Other Names: Relugolix Combination Therapy (Rel-CT); Myfembree
  Arms: Rel-CT

SUMMARY:
The goal of this investigator-initiated single-site clinical trial is to compare the overall quality of life of participants taking Relugolix combination therapy (Rel-CT) following excisional surgery for endometriosis to participants that do not take Rel-CT following the same surgery. Rel-CT is an FDA approved form of medical treatment for endometriosis. It is known to work in treating endometriosis pain. However, investigators do not know whether or not there is a benefit to beginning Rel-CT immediately following surgery. This study will test if patients who take Rel-CT after surgery have better quality of life and less chance the endometriosis comes back, requiring additional surgery.

The main question it aims to answer is:

- Does taking Rel-CT following excisional surgery for endometriosis result in higher Endometriosis Health Profile 30 (EHP-30) scores, indicating a positive impact on overall health-related quality of life and well-being?

Participants will:

* Be randomly assigned to one of two treatment groups. One treatment group will take study drug Rel-CT after having excisional surgery, and the other treatment group will just have the surgery alone.
* Be asked to complete questionnaires, called the Endometriosis Health Profile 30 (EHP-30) at 4 timepoints. The first time is before surgery, then at follow-up visits at 1 month, 3 months, and 6 months. The survey has 30 questions that ask about pain, control, powerlessness, emotional well-being, social support, and self-image.

Researchers will compare the two treatment groups (Rel-CT and non Rel-CT) to see if there is a change in EHP-30 scores.

DETAILED DESCRIPTION:
The design of this study will be an unblinded randomized controlled trial of medical suppression with once daily Relugolix combination therapy (Rel-CT) following excisional surgery for endometriosis performed by high volume minimally invasive gynecologic surgeons. Women over the age of 18 scheduled to undergo a laparoscopic surgery for endometriosis will be screened and if agree and consented to participate will be randomized to either Rel-CT following surgery or no post-operative hormonal suppression using a block randomization with blocks 2 and 4. The surgeon will not have access to the randomization schedule to reduce selection bias. Inclusion criteria will include: 1) Patients over the age of 18 planning to undergo an elective laparoscopic/robotic procedure for known or suspected endometriosis. Exclusion criteria will include: 1) Patients with known contraindications to REL-CT; 2) Any form of hormonal suppression of endometriosis within the protocol guidelines; 3) Primary language other than English/Spanish; 4) Patients without histologic evidence of endometriosis following their surgical procedure; 5) Patients interested in pregnancy within the 12 months following their surgical procedure.

The primary outcome will be change in Endometriosis Health Profile 30 (EHP-30) score. A preoperative EHP-30 will be completed by all patients enrolled in the study within 4 weeks of their scheduled surgical procedure and then again postoperatively at 1 month, 3 months, and 6 months. Investigators expect that postoperative use of REL-CT will lead to a clinically meaningful improvement in EHP-30 scores compared to surgery alone. In addition, investigators will gather data on our secondary outcomes: These data could be very helpful in informing providers and patients of the utility of medical suppression of endometriosis using REL-CT following surgery.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Planning to undergo an elective laparoscopic or robotic procedure for known or suspected endometriosis

Exclusion criteria

-A known contraindication to REL-CT. Contraindications include:

* High risk of arterial, venous thrombotic, or thromboembolic disorder
* Pregnancy Known osteoporosis
* Current or history of breast cancer or other hormone-sensitive malignancies
* Known hepatic impairment or disease
* Undiagnosed abnormal uterine bleeding
* Known hypersensitivity to components of Rel-CT
* The patient did not discontinue hormonal suppression within the required timeline:

Trans-Dermal, Oral Medication, Patch, or Vaginal Ring: day before surgery

Intrauterine Device or Sub-Dermal Implant: removed at surgery

Injectable Medication: at least 12 weeks before surgery

* Primary language other than English/Spanish
* Interested in pregnancy within the 6 months following the surgical procedure.
* If pregnancy test performed during pre-surgical work up is positive, the patient will no longer be a candidate for endometriosis surgery and will therefore not be eligible for the study.
* Patients without histologic evidence of endometriosis following their surgical procedure will be removed from the study prior to receiving the study intervention.
* Patients who undergo a surgical intervention more invasive than the planned laparoscopic or robotic excisional surgery, such as open abdominal surgical repair, will be removed from the study prior to receiving the study intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biological female at birth and meeting criteria for endometriosis
Enrollment: 110 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
This study aims to determine if immediate postoperative medical suppression with Regugolix combination therapy (Rel-CT) following excisional surgery for endometriosis is superior to surgery alone. | 6 months
  The study will assess quality of life via change in total Endometriosis Health Profile 30 (EHP-30) scores following excisional surgery for endometriosis from baseline to 6 months postoperatively.

SECONDARY OUTCOMES:
Change in EHP-30 scores between groups stratified by endometriosis stage | 6 months
  Comparison of EHP-30 scores according to endometriosis stage of the participant of Rel-CT group to non Rel-Ct treatment group
Comparison of EHP-30 subscales | 6 months
  Comparison of EHP-30 survey subscales in treatment groups.
Comparison of EHP-30 by superficial vs deep infiltrating types | 6 months
  Comparison of EHP-30 scores according to the participant having superficial or deep infiltrating endometriosis post-surgery.
Reintervention rates between groups | 6 months
  Need for surgical reintervention will be assessed between treatment groups.
Compliance rates for the study drug and office visits following surgery | 6 months
  Study drug adherence will be monitored and reported.
Rates of concomitant adenomyosis | 6 months
  Rate of concomitant adenomyosis will be collected and compared between two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Klebanoff, MD, Principal Investigator — Main Line Health
Locations (1):
- Main Line Health, Wynnewood, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Estimating the Mean and Variance from the Median, Range, and the Size of a Sample — https://bmcmedresmethodol.biomedcentral.com/articles/10.1186/1471-2288-5-13

DOCUMENTS (1):
  • Informed Consent Form (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT06439524/ICF_002.pdf